CLINICAL TRIAL: NCT03060226
Title: Prediction of Appearance of Late Cutaneous Side Effects After RadioTherapy
Acronym: PAESCART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A02021-50
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Merkel Carcinoma; Radiotherapy Side Effect
MeSH Terms: conditions — Radiation Injuries | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other)
  Interventions: Diagnostic Test: blood sample
- radiosensibility group (Other)
  Interventions: Diagnostic Test: blood sample

INTERVENTIONS:
Diagnostic Test: blood sample — Search of blood predictive marker (s)

SUMMARY:
Search for blood predictive marker (s) for cutaneous radiosensitivity

ELIGIBILITY:
Inclusion Criteria:

* Patient treated with surgery and radiotherapy (RT) for histologically proven Merkel carcinoma
* Previous radiotherapy treatment completed for at least 6 months
* Absence of prior treatment by chemotherapy or hormonotherapy
* Patient over 18 years of age
* Patient affiliated to a social security system
* Informed consent signed

Exclusion Criteria:

* Presence of another evolutionary cancer
* Re-irradiation in the same area
* Absence of available dosimetry data
* Patient under guardianship or curatorship or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Identification and dosage of blood predictive marker(s) | 1 blood sample at inclusion
  Concentration of IL-1α, IL-1β, IL-4, IL-6, IL-8, IL-10, TNF-α, TGF-β, IL-13, IL-17 and CRP
Identification and dosage of blood predictive marker(s) | 1 blood sample at inclusion
  Concentration of 8-OHdG extracellular, Antioxidant enzymes (catalase, superoxyde dismutase, glutathion peroxydase)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre François Baclesse, France, France

IPD SHARING:
Plan to Share IPD: No